CLINICAL TRIAL: NCT05401370
Title: Role of Methylene Blue Dye in Identification of Facial Nerve in Parotid Surgery
Brief Title: Role of Methylene Blue in Parotid Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ismail Ali Mohamed Ismail, Resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MB in parotid surgery
Record Dates: First submitted 2022-04-25; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Parotid Tumor
MeSH Terms: conditions — Parotid Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MB group (Active Comparator): Mb group will undergo surgeries with methylene blue staining
  Interventions: Procedure: Methylene blue dye
- Control group (No Intervention): Control group will undergo surgeries without methylene blue staining

INTERVENTIONS:
Procedure: Methylene blue dye — For MB group, the staining of the glandular tissue will be obtained with 3-4 mL of 1% MB that will be introduced into the gland via the salivary duct several minutes before the surgery.The trans-oral catheterization of the Stensen's duct will be performed and the solution will be injected via intravenous cannula.The glandular tissue will turn dark blue.
  Arms: MB group

SUMMARY:
usefulness of the methylene blue staining for identification of facial nerve in parotid gland surgery

DETAILED DESCRIPTION:
The specific surgical morbidity remains significant in parotid gland surgery. In addition to temporary facial weakness and permanent facial nerve injury, postparotidectomy depression and Frey's syndrome (gustatory sweating) are specific for this type of surgery. To reduce the surgical morbidity, several modifications of parotidectomy have been implemented but postsurgical complications remain especially facial nerve injury . To overcome this difficulty, an identification method might be used such as preoperative intravital staining of the gland with methylene blue (MB).

Although MB staining is not designed to be used as a sole technique, it can be combined with other techniques such as identification of the anatomic landmarks. MB staining is simple, inexpensive, and not time consuming technique.It is an indirect facial nerve identification technique, because there is no nerve handling,thus decreasing iatrogenic nerve impairment.After injection of the parotid gland with MB dye, fine white nerve fibers can be observed . Tumors in the parotid gland are also easily seen because they are not stained and will be visible in the surgical field.

ELIGIBILITY:
Inclusion Criteria:

* All new cases presented with primary benign or malignant parotid tumors.

Exclusion Criteria:

* Cases with secondary tumors of the gland

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of cases that don't develop post surgical parotidectomy facial nerve weakness after using preoperative intravital staining of the gland with methylene blue dye. | One year
  Twenty cases presented to outpatient clinic in Assiut university hospital with benign or primary malignant parotid gland tumors will be included in the study, clinically evaluated, confirmation of diagnosis will be achieved by CT, MRI, or CT/MRI investigations , ultrasonography and fine-needle aspiration biopsy (FNAB).
  then Divide the selected cases into two groups randomly; group A for surgeries with MB staining and group B for surgeries without MB staining that serves as control group. type of surgery will be chosen according to CT or MRI data and fine-needle aspiration biopsy (FNAB)then Follow up facial nerve injury manifestations for the included cases for one year for comparison between 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Ali Mohamed, Principal Investigator — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Age,sex,clinical diagnosis.
Supporting Information: Study Protocol, SAP
Time Frame: 3 years
Access Criteria: Age,sex,clinical diagnosis.